CLINICAL TRIAL: NCT01417130
Title: Alzheimer's Disease Anti-Inflammatory Prevention Trial Follow-Up Study
Brief Title: Follow-up Study of the Alzheimer's Disease Anti-Inflammatory Prevention Trial
Acronym: ADAPT-FS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: VA Puget Sound Health Care System (U.S. Federal Agency); National Institute on Aging (NIA) (NIH); Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: BREITNERBJ18CO; 5U01AG015477-07 (NIH)
Record Dates: First submitted 2011-06-24; First posted 2011-08-16 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2012-01

CONDITIONS: Alzheimer Disease; Dementia
Keywords: Naproxen; Celecoxib; Anti-Inflammatory Agents, Non-Steroidal
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimens retained from the ADAPT trial include plasma, serum, urine and cerebrospinal fluid (the latter from a smaller sample of volunteers). Additional collection of cerebrospinal fluid from prior donors and from a new panel of volunteers is conducted under a different sub-study of ADAPT.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Naproxen sodium (220 mg b.i.d): Original assignment in the ADAPT trial
- Celecoxib (200 mg b.i.d.): Original assignment in the ADAPT trial
- Placebo: Original assignment in the ADAPT trial

SUMMARY:
The Alzheimer's Disease Anti-inflammatory Prevention Trial - Follow-up Study (ADAPT-FS) will continue observations of the declared primary outcomes of the Alzheimer's Disease Anti-inflammatory Prevention Trial (ADAPT) in the cohort previously established for that trial.

DETAILED DESCRIPTION:
ADAPT was a multicenter, randomized, placebo-controlled trial designed to test the safety and efficacy of naproxen and celecoxib for the primary prevention of Alzheimer's Disease (AD) dementia and for attenuation of age related cognitive decline in persons over 70 years of age. The ADAPT treatments were stopped on 17 December, 2004, after the substantial majority of participants had been given treatments over an interval of one to three years. Participants remained under observation until May, 2006, using double-masked methods of case identification that were identical to those of the original ADAPT protocol. Results from the entire period of observations in ADAPT were ambiguous and suggested a need for additional longitudinal data to learn whether the dual-inhibitor NSAID naproxen can effect a long-term reduction in the occurrence of AD dementia.

This ADAPT Follow-up Study (ADAPT-FS) is following-up the participants originally enrolled in ADAPT after a further interval of four years, thereby identifying additional individuals with AD dementia in each treatment assignment group, and then using time-dependent methods to estimate and contrast incidence rates by treatment assignment. The study is also extending prior observations on trajectory of cognitive performance on several psychometric measures, thus testing the hypothesis of differences in such trajectory by treatment assignment in ADAPT.

ADAPT-FS is sponsored by the National Institute on Aging (NIA) and is being conducted at the Roskamp Institute in Tampa, FL; the Veterans Affairs Puget Sound Health Care System in Seattle, WA; Boston University School of Medicine, in Boston, MA; the Johns Hopkins Medical Institutions, in Baltimore, MD; Sun Health Research Institute, in Phoenix, AZ; and the University of Rochester, in Rochester, NY.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have been enrolled previously in the Alzheimer's Disease Anti-Inflammatory Prevention Trial (ADAPT).

Exclusion Criteria:

* Individuals not previously enrolled in the ADAPT trial.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Living members of the cohort previously enrolled in the Alzheimer's Disease Anti-inflammatory Prevention Trial (ADAPT)
Sampling Method: Non-Probability Sample
Enrollment: 1650 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-10 (Actual); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Incident Alzheimer's Disease dementia | Up to 9 years.
  Incidence

SECONDARY OUTCOMES:
Trajectory of performance on cognitive tests in relation to ADAPT treatment assignment | Up to 9 years.
  Telephone Interview for Cognitive Status (TICS), Rivermead Behavioral Memory Test (RBMT), Generative Verbal Fluency (GVF)

CONTACTS AND LOCATIONS:
Overall Officials: John CS Breitner, MD, MPH, Study Chair — Veteran Affairs Puget Sound Health Care System; Laura D Baker, PhD, Study Director — Veteran Affairs Puget Sound Health Care System; Constantine Lyketsos, MD, MHS, Principal Investigator — The Johns Hopkins University; Peter Zandi, PhD, Principal Investigator — The Johns Hopkins University; Denis Evans, MD, Principal Investigator — Rush Institute for Healthy Aging
Locations (6):
- United States (6):
  - Banner Sun Health Research Institute, Sun City, Arizona
  - The Roskamp Institute, Sarasota, Florida
  - The Johns Hopkins University, Baltimore, Maryland
  - Boston University School of Medicine, Boston, Massachusetts
  - Monroe Community Hospital, Rochester, New York
  - Veterans Affairs Puget Sound Health Care System, Seattle, Washington

REFERENCES:
- [Background] ADAPT Research Group; Lyketsos CG, Breitner JC, Green RC, Martin BK, Meinert C, Piantadosi S, Sabbagh M. Naproxen and celecoxib do not prevent AD in early results from a randomized controlled trial. Neurology. 2007 May 22;68(21):1800-8. doi: 10.1212/01.wnl.0000260269.93245.d2. Epub 2007 Apr 25. PMID 17460158
- [Background] ADAPT Research Group. Cardiovascular and cerebrovascular events in the randomized, controlled Alzheimer's Disease Anti-Inflammatory Prevention Trial (ADAPT). PLoS Clin Trials. 2006 Nov 17;1(7):e33. doi: 10.1371/journal.pctr.0010033. PMID 17111043
- [Background] ADAPT Research Group; Martin BK, Szekely C, Brandt J, Piantadosi S, Breitner JC, Craft S, Evans D, Green R, Mullan M. Cognitive function over time in the Alzheimer's Disease Anti-inflammatory Prevention Trial (ADAPT): results of a randomized, controlled trial of naproxen and celecoxib. Arch Neurol. 2008 Jul;65(7):896-905. doi: 10.1001/archneur.2008.65.7.nct70006. Epub 2008 May 12. PMID 18474729
- [Background] Meinert CL, Martin BK, McCaffrey LD, Breitner JC. Do we need to adjudicate major clinical events? Clin Trials. 2008;5(5):557; author reply 558. doi: 10.1177/1740774508096007. No abstract available. PMID 18827048
- [Background] Martin BK, Breitner JC, Evans D, Lyketsos CG, Meinert CL. The trialist, meta-analyst, and journal editor: lessons from ADAPT. Am J Med. 2007 Mar;120(3):192-3. doi: 10.1016/j.amjmed.2006.12.010. No abstract available. PMID 17349436
- [Background] Breitner J, Evans D, Lyketsos C, Martin B, Meinert C. ADAPT trial data. Am J Med. 2007 Mar;120(3):e3; author reply e5; discussion e7. doi: 10.1016/j.amjmed.2006.09.022. No abstract available. PMID 17349430
- [Background] Breitner JC, Martin BK, Meinert CL. The suspension of treatments in ADAPT: concerns beyond the cardiovascular safety of celecoxib or naproxen. PLoS Clin Trials. 2006 Dec 22;1(8):e41. doi: 10.1371/journal.pctr.0010041. No abstract available. PMID 17192795
- [Background] Martin BK, Meinert CL, Breitner JC; ADAPT Research Group. Double placebo design in a prevention trial for Alzheimer's disease. Control Clin Trials. 2002 Feb;23(1):93-9. doi: 10.1016/s0197-2456(01)00189-1. PMID 11852171
- [Derived] ADAPT-FS Research Group. Follow-up evaluation of cognitive function in the randomized Alzheimer's Disease Anti-inflammatory Prevention Trial and its Follow-up Study. Alzheimers Dement. 2015 Feb;11(2):216-25.e1. doi: 10.1016/j.jalz.2014.03.009. Epub 2014 Jul 9. PMID 25022541
- See also: Alzheimer's Disease Anti-Inflammatory Prevention Trial — http://clinicaltrials.gov/ct2/show/NCT00007189